CLINICAL TRIAL: NCT04581525
Title: Modulating Neuropathic Pain With Transcranial Direct Current Stimulation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient staff to carry out study
Sponsor: Susan McDowell (Other)
Collaborators: Foundation for Physical Medicine and Rehabilitation (Other)
Responsible Party: Sponsor-Investigator, Susan McDowell, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 45535
Record Dates: First submitted 2020-09-28; First posted 2020-10-09 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Pain, Neuropathic; Complex Regional Pain Syndromes; Phantom Limb Pain; Spinal Cord Injuries
Keywords: neuroplasticity; rehabilitation; transcranial direct current stimulation
MeSH Terms: conditions — Neuralgia; Complex Regional Pain Syndromes; Phantom Limb; Spinal Cord Injuries | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tDCS of DLPFC (Experimental): Subjects will receive 20 minutes of active transcranial direct current stimulation at 2mA applied to the left dorsolateral prefrontal cortex (DLPFC). Subjects will undergo stimulation once a day for 10 consecutive weekdays.
  Interventions: Device: transcranial direct current stimulation
- tDCS of M1 (Experimental): Subjects will receive 20 minutes of active transcranial direct current stimulation at 2mA applied to the left primary motor cortex (M1). Subjects will undergo stimulation once a day for 10 consecutive weekdays.
  Interventions: Device: transcranial direct current stimulation
- Sham tDCS (Sham Comparator): Subjects will receive 20 minutes of sham transcranial direct current stimulation. Subjects will undergo stimulation once a day for 10 consecutive weekdays.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation

SUMMARY:
This study will examine whether a form of non-invasive brain stimulation can help reduce pain in people with persistent neuropathic pain.

DETAILED DESCRIPTION:
This study will look at the effects of a painless, non-invasive form of brain stimulation, called transcranial direct current stimulation, or tDCS. tDCS is thought to increase the brain's ability to change. Participants will be assigned to one of three groups by chance. Two groups will receive tDCS at a level expected to increase the brain's ability to change, while the other group will receive tDCS at a level not thought to affect the brain's ability to change.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Have chronic (>12 months) neuropathic pain, including but not limited to complex regional pain syndrome, phantom limb pain, or pain of neurogenic origin following spinal cord injury

Exclusion Criteria:

* History of seizures or epilepsy
* Addition or change in the dosage of drugs now to interfere with pain within 1 month of enrollment
* Untreated depression
* History of head injury with loss of consciousness, severe alcohol or drug abuse, or psychiatric illness
* Positive pregnancy test or being of childbearing age and not using appropriate contraception
* Presence of ferromagnetic material in the cranium except in the mouth, including metal fragments from occupational exposure, and surgical clips in or near the brain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-06-07 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
Change in McGill Pain Questionnaire from baseline 1 and 2 average | Baseline 1: 1 week before starting intervention, Baseline 2: immediately before starting intervention, Intervention mid-point: after 5 days intervention, Post-intervention: after 10 days intervention, Follow up: 1 month after completing intervention
  This self-reported assessment measures intensity and quality of pain. Scores can range from 0 to 45. A decrease in score indicates an improvement in pain.

SECONDARY OUTCOMES:
Change in Short-Form 36 Health Survey from baseline 1 and 2 average | Baseline 1: 1 week before starting intervention, Baseline 2: immediately before starting intervention, Intervention mid-point: after 5 days intervention, Post-intervention: after 10 days intervention, Follow up: 1 month after completing intervention
  This self-reported assessment provides information regarding an individual's perception of their health and quality of life. Scores range from 0 to 100. An increase in score indicates an improvement in perceived health and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Susan McDowell, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky at Cardinal Hill Rehabilitation Hospital, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No